CLINICAL TRIAL: NCT05514743
Title: Response of Cardiovascular Parameters to Physical Therapy Post Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Omnia Saeed Mahmoud Ahmed, Dr.Omnia Saeed Mahmoud Ahmed, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: HS000107
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Liver Transplant; Complications
MeSH Terms: interventions — Blood Pressure Monitors

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart rate (Active Comparator): Heart rate monitors can assess a person's heart rate and reveal whether it is high or low. Heart rate Trusted Source is a "clinical indicator of overall cardiac health," and it can also help a person determine their performance during a workout.
  Interventions: Procedure: 6 minute walk test , Blood pressure monitoring
- Blood pressure (Active Comparator): It will be carried out before and after interventions to determine the patients functional capacity (in the 7th.day &in the 21st.day.) It will be used as a training tool as well as an assessment tool.
  Interventions: Procedure: 6 minute walk test , Blood pressure monitoring

INTERVENTIONS:
Procedure: 6 minute walk test , Blood pressure monitoring — Heart rate monitors can assess a person's heart rate and reveal whether it is high or low. Heart rate Trusted Source is a "clinical indicator of overall cardiac health," and it can also help a person determine their performance during a workout.
  Six minute walk test:
  It will be carried out before and after interventions to determine the patients functional capacity (in the 7th.day &in the 21st.day.) It will be used as a training tool as well as an assessment tool. They will receive conventional physical therapy program which includes deep breathing exercise in form of (diaphragmatic, apical and costal breathing), Training about right way of cough and early ambulation from bed for 3 sessions / week, twice daily for 21 days.

SUMMARY:
Liver transplantation (LT) is the only life-saving treatment option in patients with advanced liver disease. Deceased-donor LT is not frequent but is increasing in Asian countries. Because current liver allocation policies follow the severity principle wherein patients at highest risk for mortality receive top priority, anesthesiologists may face severely ill patients more frequently with deceased-donor LT than with living-donor LT. In this regard, with the outstanding surgical success of recent LT, cardiovascular complications have emerged as the leading cause of death after LT, particularly among those with advanced liver cirrhosis

DETAILED DESCRIPTION:
Cardiovascular complications have emerged as the leading cause of death after liver transplantation, particularly among those with advanced liver cirrhosis. Therefore, a thorough and accurate cardiovascular evaluation with clear comprehension of cirrhotic cardiomyopathy is recommended for optimal anesthetic management. However, cirrhotic patients manifest cardiac dysfunction concomitant with pronounced systemic hemodynamic changes, characterized by hyperdynamic circulation such as increased cardiac output, high heart rate, and decreased systemic vascular resistance. These unique features mask significant manifestations of cardiac dysfunction at rest, which makes it difficult to accurately evaluate cardiovascular status As cardiovascular complications are leading causes of nongraft related mortality after LT [2], the importance of identifying masked intrinsic cardiac dysfunction or decreased capacity of cardiac contractility due to external stress has been emphasized. However, detecting ventricular dysfunction in a resting state is difficult, as marked vasodilation and increased arterial compliance lead to latent or mild cardiac manifestations [4]. Different stress tests, using drugs or exercise, have been applied to unmask cardiac dysfunction; however, achieving a target HR and blood pressure is difficult given the poor functional conditions of patients with LC [5].

Dobutamine stress echocardiography (DSE) is recommended to discriminate high-risk patients with ischemic heart disease; however, the accuracy of DSE varies widely among studies as a result of various selection criteria [3] and the inability to achieve the predicted target HR to provoke wall motion abnormalities. This inadequacy is based on the failure of beta receptors to respond to sympathetic stimulation in patients with LC or the use of beta blockers to prevent variceal bleeding. Therefore, the accuracy of DSE is questionable, and its sensitivity is reported as low as 13-14% [6-7]. Nicolau-Raducu et al. [8] demonstrated that DSE has 9% sensitivity, 33% positive predictive value, and 89% negative predictive value for predicting early cardiac events after LT.

The autonomic nervous system is an important regulator of cardiovascular homeostasis, and an HR analysis is considered a surrogate of vagal and sympathetic disturbances. Therefore, HR measurements have been recognized as a prognostic factor in many clinical investigations [9-12]. Studies showing reduced HR variability, which correlates with disease severity, central hypovolemia, and the degree of portal hypertension have also been reported [13-14]. Kim et al. [15] found that sympathetic withdrawal is associated with hypotension after graft reperfusion during LT.

Patients with LC have an increased resting HR due to hyperdynamic circulation, increased circulating catecholamines, and cirrhotic cardiomyopathy [16-17]. Kwon et al. [18] demonstrated that resting HR is associated with all-cause mortality in LT recipients and showed that patients with HR >80 beats/min are significantly associated with a higher risk for all-cause mortality (hazard ratio 1.83) compared to patients with HR ≤65 beats/min.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 40 to 60
2. All patients will be medically stable.
3. All patients will have the same medical care (fluid and electrolyte management in the ICU, immunosuppressive, prophylactic) the patient might also require (antihypertensive medications, insulin or oral hypoglycemic agents, mild analgesics).

Exclusion Criteria:

* All patients will be subjected to full clinical history and full clinical examination for exclusion of the following:

  1. Patients with neurological and neuromuscular disease.
  2. Total liver transplantation.
  3. Cardiac disease.
  4. Alcoholic hepatitis.
  5. Blind individuals.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | 3 weeks
  Heart rate monitors can assess a person's heart rate and reveal whether it is high or low. Heart rate Trusted Source is a "clinical indicator of overall cardiac health," and it can also help a person determine their performance during a workout.
  Six minute walk test:
  It will be carried out before and after interventions to determine the patients functional capacity (in the 7th.day &in the 21st.day.) It will be used as a training tool as well as an assessment tool.
Blood pressure | 3 weeks
  It will be carried out before and after interventions to determine the patients functional capacity (in the 7th.day &in the 21st.day.) It will be used as a training tool as well as an assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Omnia Saeed, PhD, Principal Investigator — October University for Modern Sciences and Arts
Locations (1):
- El Sahel Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watt KD, Pedersen RA, Kremers WK, Heimbach JK, Charlton MR. Evolution of causes and risk factors for mortality post-liver transplant: results of the NIDDK long-term follow-up study. Am J Transplant. 2010 Jun;10(6):1420-7. doi: 10.1111/j.1600-6143.2010.03126.x. Epub 2010 May 10. PMID 20486907
- [Background] Zaky A, Bendjelid K. Appraising cardiac dysfunction in liver transplantation: an ongoing challenge. Liver Int. 2015 Jan;35(1):12-29. doi: 10.1111/liv.12582. Epub 2014 Jun 5. PMID 24797833
- [Background] Wong F, Liu P, Lilly L, Bomzon A, Blendis L. Role of cardiac structural and functional abnormalities in the pathogenesis of hyperdynamic circulation and renal sodium retention in cirrhosis. Clin Sci (Lond). 1999 Sep;97(3):259-67. PMID 10464050
- [Background] Kwon HM, Jun IG, Jung KW, Moon YJ, Shin WJ, Song JG, Hwang GS. Pretransplant Resting Heart Rate and Its Association With All-Cause Mortality in Liver Transplant Recipients. Transplant Proc. 2017 Jun;49(5):1092-1096. doi: 10.1016/j.transproceed.2017.03.043. PMID 28583534
- See also: Cardiovascular dysfunction and liver transplantation. Korean journal of anesthesiology, 71(2), 85-91. — https://doi.org/10.4097/kjae.2018.71.2.85